CLINICAL TRIAL: NCT04883905
Title: ELEVATE, a Global Observational Longitudinal Prospective Registry of Patients With Acute Hepatic Porphyria (AHP)
Brief Title: ELEVATE, a Registry of Patients With Acute Hepatic Porphyria (AHP)
Acronym: ELEVATE
Status: Recruiting | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-AS1-006; EUPAS43201 (Registry Identifier: EU PAS REGISTER)
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Hepatic Porphyria
Keywords: Givosiran; AHP; Acute hepatic porphyria
MeSH Terms: conditions — Coproporphyria, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with AHP: Patients with a diagnosis of AHP will be eligible for the study and will be managed and treated per routine clinical practice.

SUMMARY:
This global patient registry is being conducted to characterize the natural history and real-world clinical management of patients with AHP, and to further characterize the real-world safety and effectiveness of givosiran and other approved AHP therapies.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of AHP, per physician's determination

Exclusion Criteria:

* Currently enrolled in a clinical trial for any investigational agent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with all types of AHP, including patients with hepatic and/or renal impairment, adolescents, elderly patient, and pregnant or lactating women.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Selected Events of Interest in AHP Patients | Up to 6 years
  Selected events of interest are defined as hepatic events (including hepatic neoplasia), renal events, thromboembolic events, and pancreatitis.

SECONDARY OUTCOMES:
Annualized Rate of Porphyria Attacks | Up to 6 years
  Porphyria attacks are defined as meeting all of the following criteria: an acute episode of neurovisceral pain in the abdomen, back, chest, extremities and/or limbs, no other medically determined cause, and requires treatment with intravenous (IV) dextrose or hemin, carbohydrates, or analgesics, or other medications such as antiemetics at a dose or frequency beyond the participant's usual daily porphyria management.
12-Item Short Form Health Survey Version 2 (SF-12 V2) (Standard Version) | Up to 6 years
  S-12 V2 is a 12-question measure capturing global quality of life and overall health status and evaluates the following 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (29):
- United States (13):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, Gilbert, Arizona
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Minneapolis, Minnesota
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Oklahoma City, Oklahoma
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Galveston, Texas
  - Clinical Trial Site, Salt Lake City, Utah
  - Clinical Trial Site, Seattle, Washington
- Clinical Trial Site, Leuven, Belgium
- France (3):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Paris
  - Clinical Trial Site, Toulouse
- Germany (3):
  - Clinical Trial Site, Berlin
  - Clinical Trial Site, Chemnitz
  - Clinical Trial Site, Würzburg
- Italy (2):
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Modena
- Clinical Trial Site, Madrid, Spain
- Clinical Trial Site, Stockholm, Sweden
- Clinical Trial Site, Zurich, Switzerland
- Taiwan (2):
  - Clinical Trial Site, Taichung
  - Clinical Trial Site, Taipei
- United Kingdom (2):
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No